CLINICAL TRIAL: NCT00798395
Title: A Randomized Double-blind, Placebo-controlled, 4-period Cross-over Study to Assess the Effect of Single and Multiple Doses of 1.5 mg and 4.5 mg Org 50081 and a Single Dose of 7.5 mg Zopiclone on Next-day Driving Ability and Psychomotor Performance in Healthy Volunteers.
Brief Title: A Study to Assess the Effect of Single and Multiple Doses Org 50081 and a Single Dose of Zopiclone on Next-day Driving Ability and Psychomotor Performance in Healthy Volunteers. (P05794) (COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P05794; 21105
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Sleep Initiation and Maintenance Disorders; Mental Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Mental Disorders | interventions — Mirtazapine; zopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment 1 (Experimental)
  Interventions: Drug: Org 50081
- Treatment 2 (Experimental)
  Interventions: Drug: Org 50081
- Treatment 3 (Placebo Comparator)
  Interventions: Drug: Placebo
- Treatment 4 (Active Comparator)
  Interventions: Drug: zopiclone

INTERVENTIONS:
Drug: Org 50081 — 1.5 mg on day 1-7
  Arms: Treatment 1
Drug: Org 50081 — 4.5 mg on Day 1-7
  Arms: Treatment 2
Drug: Placebo — Once daily on Day 1-7
  Arms: Treatment 3
Drug: zopiclone — Single dose of 7.5 mg
  Arms: Treatment 4

SUMMARY:
This trial is to investigate the effect on next-day driving performance and psychomotor performance in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject has at least 3 years of car driving experience
* Subject signs the trial Informed Consent Form
* Subject is in a healthy condition as judged by the investigator
* Subject has a regular sleep pattern

Exclusion Criteria:

* Subject has insomnia or any other sleep disorder
* Medication or drug use of any kind prior to the study
* Relevant history or presence of a significant medical illness

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The Standard Deviation of Lateral Position | Day 8

SECONDARY OUTCOMES:
Psychomotor and cognitive performance tasks | Day 8